CLINICAL TRIAL: NCT03513770
Title: Autonomic Control of the Circulation and the Venous Distension Reflex
Brief Title: Autonomic Control of the Circulation and VDR
Acronym: VDR
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jian Cui, Associate Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00006585
Record Dates: First submitted 2018-02-15; First posted 2018-05-02 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Venous Distension Reflex; Blood Pressure
MeSH Terms: interventions — Salicylic Acid; Ketorolac Tromethamine

STUDY DESIGN:
Intervention Model Description: The investigators will examine (using a prospective observational design) if a COX blockade will inhibit the Muscle Sympathetic Nerve Activity response to venous distension, and if a COX blockade will alter vein sizes during venous distension using MRI. Each subject will serve as their own control.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: These two trials (A and B) will be performed in random order and in a doubleblind fashion for subjects and the data analyzing team. The medical staff who prepare and administrate the drugs and monitor the subject's safety, will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac (Experimental): The Wrist-to-Elbow occlusion procedure will be performed followed by 2 ketorolac tromethamine + saline infusions into the occluded arm.
  Interventions: Other: Wrist-to-elbow (W-E) occlusion; Drug: ketorolac tromethamine
- Control (Placebo Comparator): The Wrist-to-Elbow occlusion procedure will be performed followed by 2 saline only infusions into the occluded arm.
  Interventions: Other: Wrist-to-elbow (W-E) occlusion; Drug: saline control

INTERVENTIONS:
Other: Wrist-to-elbow (W-E) occlusion — An IV will be inserted in the antecubital fossa of one arm. The arm will be fitted with occlusion cuffs arranged in a continuous fashion from the wrist to the elbow. A final cuff will be placed on the upper arm. The cuffs from the wrist to the elbow will be inflated to the same pressure of up to 300 mmHg using a pressurized air tank.
  First, the subject?s arm will be elevated and the subject will make a fist to squeeze blood from the hand. Then the wrist cuff will be inflated. Once that cuff is fully inflated, the next cuff in the sequence will be inflated. Cuffs are inflated in sequence until the elbow cuff is inflated. After a 10-15 second period to allow blood to drain, the upper arm cuff will inflate (up to 250 mmHg) to keep any additional blood from entering the forearm. Next, the cuffs on the forearm will be removed but the upper arm cuff will remain inflated.
Drug: ketorolac tromethamine — In the COX blockade trial, just after the Wrist-to-elbow occlusion, 6 mg ketorolac tromethamine in 10 ml saline will be infused into the forearm over 1 minute. After 10 minutes, a second infusion of ketorolac tromethamine (up to 3 mg) in 5% of the forearm volume of saline,( ~40-60 ml) will be infused into the occluded forearm at a rate of ~ 30 ml/min. Five minutes of data will then be collected before releasing the upper arm cuff. Infusion 1 is to block the COX pathway, while infusion 2 is to induce venous distension.
  Arms: Ketorolac
Drug: saline control — In the saline control trial performed on a separate day, saline (without ketorolac) in identical volumes as those in the COX blockade trial, will be infused.
  Arms: Control

SUMMARY:
The study objective of this project is to examine the mechanisms of the venous distension reflex (VDR) in humans. We hypothesize that COX blockade with ketorolac tromethamine, an intravenous NSAID, will attenuate the muscle sympathetic nerve activity (MSNA) response to limb venous distension. To gain further insight into whether the COX byproducts directly stimulate chemically-sensitive afferents, or enable venodilation and indirectly evoke afferent stimulation, we will measure vein size using 3T MRI during venous distention with and without ketorolac infusions.

DETAILED DESCRIPTION:
We will use a prospective observational design to examine if a COX blockade will inhibit the MSNA response to venous distension (Aim1), and if a COX blockade will alter vein sizes during venous distension (Aim2). Each subject will serve as their own control.

Aim 1:

An IV will be inserted in the antecubital fossa of one arm, and the wrist-to-elbow occlusion will be performed.

To block the COX system, 6 mg ketorolac tromethamine in 10 ml saline will be infused into the forearm over 1 minute (Infusion 1). After 10 minutes, a second infusion of ketorolac tromethamine (up to 3 mg) in 5% of the forearm volume of saline,( ~40-60 ml) will be infused into the occluded forearm at a rate of ~ 30 ml/min (Infusion 2). Five minutes of data will then be collected before releasing the upper arm cuff. Infusion 1 is to block the COX pathway, while infusion 2 is to induce venous distension.

In the saline control trial, saline (without ketorolac) in identical volumes as those in the COX blockade trial will be performed on a separate day.

Aim 2:

The subject will lie supine inside the MRI scanner. The subject will be instrumented with cuffs for the wrist-to-elbow occlusion procedure on one arm, and cuffs for automated BP and HR measurements from the other arm, The images will be obtained before and during the wrist-to-elbow occlusion procedure. The sizes of veins (i.e. cross sectional area) will be measured offline.

ELIGIBILITY:
Inclusion Criteria

* Are capable of giving informed consent
* Are any race or ethnicity
* Are fluent in written and spoken English
* Have a satisfactory history and physical exam to meet inclusion/exclusion criteria
* Are free of acute or chronic medical conditions
* Are 21 - 35 years of age (inclusive)
* Weigh over 50 kg

Exclusion Criteria

* Are less than 21 or over 35 years of age
* Are Pregnant or nursing women
* Are prisoners or institutionalized individuals or unable to consent
* Any chronic diseases (hypertension, heart, lung, neuromuscular disease, kidney disease, diabetes or cancer).
* Are taking medications that may affect their cardiovascular or nervous system
* Has taken an NSAID within 48 hours of any visit (visit will need to be rescheduled)
* Has never taken NSAIDs and therefore would not know if they are allergic to it
* Have a supine BP >140/90 mmHg
* Have known allergy to ibuprofen-like drugs (NSAIDS) or aspirin
* Have history of asthma or nasal polyps
* Have history of GI bleeding or ulcers
* Subjects with ferromagnetic metal implants
* Subjects who are claustrophobic

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-08-14 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Microneurography (MSNA) | Recorded continuously during the 3-4 hour study visit
  This technique provides direct recordings of sympathetic nerve activity directed to blood vessels in skeletal muscle and will be our primary index of sympathoexcitation. This procedure may be performed in the either leg. External mapping of the peroneal or tibial nerve course (10-60 volts, 1-5msec, 1Hz) will be performed just behind the fibular head of the leg or in the popliteal fossa. A reference electrode will be placed subcutaneously about 2-3 cm away from the recording site. Multiunit recordings of MSNA in the leg will be obtained by transcutaneous placement of a tungsten microelectrode (insulated 200 ?m diameter with a tapered un-insulated 1-5 ?m tip) into C-fiber containing fascicle in the nerve. The electrode will be manipulated to yield a neurogram with characteristic bursts of MSNA, that will be amplified, filtered, rectified and integrated to obtain a mean voltage neurogram. Analysis consists of counting burst frequency and amplitude.
Vein size with MRI | Recorded continuously during the 3-4 hour study visit
  Forearm cross sectional images will be obtained in HMC MRI facility. The proton weighted images will be obtained with Siemens Magnetom Trio 3T scanner (Siemens Medical Solutions, Erlangen, Germany). Contrast agents are not required for this completely noninvasive technique. The subject will lie supine inside the MRI scanner, and will be instrumented with an cuffs for the wrist-to-elbow occlusion procedure on one arm, and cuffs for automated BP and HR measurements from the other arm, The images will be obtained before and during the wrist-to-elbow occlusion procedure. The sizes of veins (i.e. cross sectional area) will be measured offline.

SECONDARY OUTCOMES:
Heart Rate | Recorded continuously during the 3-4 hour study visit
  Heart rate will be continuously monitored using EKG patch electrodes and monitor (Cardiocap, Datex-Ohmeda, GE Healthcare).
Blood Pressure | Recorded continuously during the 3-4 hour study visit
  Systolic and diastolic blood pressure will be monitored using an automatic, non-invasive arm cuff (SureSigns VS3, Philips, Philips Medical Systems), and on the finger with a Finometer (Finapres Medical Systems). Baseline Finometer BP will be adjusted to match the arm cuff BP.
Laser-Doppler flowmetry | Recorded continuously during the 3-4 hour study visit
  Skin blood flow will be monitored non-invasively by laser-Doppler flowmetry using special probes taped to the skin. The skin blood flow may be measured from both arms, and legs (up to 4 probes total).
Strain gauge | Recorded continuously during the 3-4 hour study visit
  The circumference changes of the forearm will be measured with strain gauges (up to 4 gauges on one arm).
Impedance | Recorded continuously during the 3-4 hour study visit
  The electrical impedance or resistance (Zo, in ohms) of a limb segment will be measured, which reflects the total fluid content of the limb. Fluid is an excellent conductor of electricity and the electrical current travels more easily through a ?wet? limb with more blood/fluid volume in the limb. The relative change in Zo will be used as an index for the fluid/blood volume change in a limb segment. By placing 2 pieces of tape with metal strips on the limb, we are able to measure impedance of the limb segment between the tapes.

OTHER OUTCOMES:
Forearm volume | Baseline
  Forearm volume will be measured by the water displacement method. The arm will be placed in the water bath up to the elbow. The baseline limb circumference will also be measured with a tape measure.
Biochemistry | 3 blood draws during the 3-4 hour study visit.
  Venous blood samples will be drawn for Thromboxane B2 (TXB2) which will be used as an index for COX blockade, and will be measured in the Pathology laboratory in Hershey Medical Center.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States